CLINICAL TRIAL: NCT02048410
Title: Efficacy of a New Symbiotic Formulation in Children With Familial Hypercholesterolemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD,pHd, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9/14
Record Dates: First submitted 2014-01-24; First posted 2014-01-29 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Dyslipidemia; Familial Hypercholesterolemia
MeSH Terms: conditions — Dyslipidemias; Hyperlipoproteinemia Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- diet plus Lactobacillus paracasei B21060 (Active Comparator): low saturated fats diet plus the symbiotic (2.5×109cfu, bid)
  Interventions: Dietary Supplement: Lactobacillus paracasei B21060; Other: low satured diet
- low saturated fats diet (Placebo Comparator): low saturated fats diet
  Interventions: Other: low satured diet

INTERVENTIONS:
Dietary Supplement: Lactobacillus paracasei B21060 — combination of probiotic (Lactobacillus paracasei B21060) and prebiotics (arabinogalactans, xyloooligosaccarides) and amine (L-glutamine)
  Arms: diet plus Lactobacillus paracasei B21060
Other: low satured diet

SUMMARY:
Probiotics have been proposed for the treatment of dyslipidemia. the investigators aimed to evaluate efficacy, tolerability and safety of a new symbiotic formulation containing a combination of probiotic and prebiotics and amine in the treatment of children affected by familial hypercholesterolemia (FH).

DETAILED DESCRIPTION:
FH subjects, aged 6-12 years, consecutively observed a Tertiary Center for Pediatric Nutrition were randomly allocated to two groups of intervention for 6 months: active group, received a low saturated fats diet plus the symbiotic (2.5×109cfu, bid) for 6 months; control group, received low saturated fats diet alone. All children received written indications for low saturated fats diet. The plasmatic lipid profile was assessed by peripheral blood sampling at T0 and T1.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 6 and ≤ 12 years.
* Diagnosis of hypercholesterolemia (LDL cholesterol> 140 mg / dl)
* Each patient must have shown resistance to dietary therapy lasting at least 6-12 months.

Exclusion Criteria:

* Age <6 or> 12 years.
* Patients undergoing drug treatment for hypercholesterolemia.
* Any medical condition that may interfere with participation in this study
* Participation in clinical trials still in progress.
* Taking pre / probiotics for more than 7 days in the 6 months prior to enrollment

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
change of LDL cholesterol after 6 months of treatment wiyh symbiotic | The plasmatic lipid profile was assessed by peripheral blood sampling at enrollment and after 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto berni canani, MD,Phd, Principal Investigator — university of naples federicoII